CLINICAL TRIAL: NCT05844449
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Efficacy of Vanzacaftor/Tezacaftor/Deutivacaftor Triple Combination Therapy in Cystic Fibrosis Subjects 1 Year of Age and Older
Brief Title: Evaluation of Long-Term Safety and Efficacy of Vanzacaftor/Tezacaftor/Deutivacaftor in Cystic Fibrosis Participants 1 Year of Age and Older
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX22-121-106; 2022-503081-74-00 (Other: EU CT)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — deutivacaftor, tezacaftor , vanzacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VNZ/TEZ/D-IVA (Experimental): Part A: Participants (Cohort 1: 6 through 11 years of age (inclusive); Cohort 2: 2 through 5 years of age (inclusive) and Cohort 3: 1 to less than (<) 2 years of age) will receive VNZ/TEZ/D-IVA once daily at doses determined based on their age and weight. The age range is based on date of informed consent in parent study.
  Part B: Participants in Cohort 1 who meet the eligibility criteria will receive VNZ/TEZ/D-IVA for an additional 96 weeks.
  Interventions: Drug: VNZ/TEZ/D-IVA

INTERVENTIONS:
Drug: VNZ/TEZ/D-IVA — Fixed-dose combination tablets or granules for oral administration.
  Other Names: VX-121/VX-661/VX-561; VX-121/VX-661/CTP-656; vanzacaftor/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability, and efficacy of vanzacaftor/tezacaftor/deutivacaftor (VNZ/TEZ/D-IVA) in participants with cystic fibrosis (CF).

ELIGIBILITY:
Key Inclusion Criteria:

Parts A and B:

• Participants who have completed study drug treatment in the parent study (VX21-121-105; NCT Number: NCT05422222)

Part B:

-Meets at least 1 of the following criteria:

* Completed study drug treatment in Part A
* Had study drug interruption(s) in Part A, but did not permanently discontinue study drug and completed study visits up to the last scheduled visit of the treatment period of Part A

Key Exclusion Criteria:

* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment, or severe hepatic impairment that might pose an additional risk in administering study drug
* History of solid organ, hematological transplantation, or cancer
* History of drug intolerance in the parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) | From Baseline up to Week 100
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) | From Baseline up to Week 196

SECONDARY OUTCOMES:
Part A (All Cohorts): Absolute Change in Sweat Chloride (SwCl) | From Baseline Through Week 96
Part B: Absolute Change in Sweat Chloride (SwCl) | From Baseline Through Week 192
Part A (Cohort 1): Absolute Change in Percent Predicted Forced Expiratory Volume (ppFEV1) | From Baseline Through Week 100
Part B: Absolute Change in Percent Predicted Forced Expiratory Volume (ppFEV1) | From Baseline Through Week 196
Part A (All Cohorts): Number of Pulmonary Exacerbation (PEx) | From Baseline Through Week 100
Part B: Number of Pulmonary Exacerbation (PEx) | From Baseline Through Week 196
Part A (All Cohorts): Number of CF- Related Hospitalizations | From Baseline Through Week 100
Part B: Number of CF- Related Hospitalizations | From Baseline Through Week 196
Part A (Cohort 1): Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain (RD) Score | From Baseline Through Week 100
Part B: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain (RD) Score | From Baseline Through Week 196
Part A (Cohorts 1 and 2): Absolute Change in Body Mass Index (BMI) | From Baseline Through Week 100
Part B: Absolute Change in Body Mass Index (BMI) | From Baseline Through Week 196
Part A (Cohorts 1 and 2): Absolute Change in BMI-for-age Z-score | From Baseline Through Week 100
Part B: Absolute Change in BMI-for-age Z-score | From Baseline Through Week 196
Part A (Cohort 3): Absolute Change in Weight-for-length | From Baseline Through Week 100
Part B: Absolute Change in Weight-for-length | From Baseline Through Week 196
Part A (Cohort 3): Absolute Change in Weight-for-length Z-score | From Baseline Through Week 100
Part B: Absolute Change in Weight-for-length Z-score | From Baseline Through Week 196
Part A (All Cohorts): Absolute Change in Weight | From Baseline Through Week 100
Part B: Absolute Change in Weight | From Baseline Through Week 196
Part A (All Cohorts): Change in Weight-for-age Z-score | From Baseline Through Week 100
Part B: Change in Weight-for-age Z-score | From Baseline Through Week 196
Part A (Cohorts 1 and 2): Absolute Change in Height | From Baseline Through Week 100
Part B: Absolute Change in Height | From Baseline Through Week 196
Part A (Cohorts 1 and 2): Absolute Change in Height-for-age Z-score | From Baseline Through Week 100
Part B: Absolute Change in Height-for-age Z-score | From Baseline Through Week 196
Part A (Cohort 3): Absolute Change in Length | From Baseline Through Week 100
Part B: Absolute Change in Length | From Baseline Through Week 196
Part A (Cohort 3): Absolute Change in Length-for-age Z-score | From Baseline Through Week 100
Part B: Absolute Change in Length-for-age Z-score | From Baseline Through Week 196

CONTACTS AND LOCATIONS:
Locations (37):
- United States (18):
  - Children's Hospital of Orange County, Orange, California
  - Stanford University - Palo Alto - Pulmonology, Palo Alto, California
  - Children's Hospital of Colorado - Pulmonology, Aurora, Colorado
  - The Emory Clinic - Clifton Road - Pulmonology, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago - Hematology, Chicago, Illinois
  - JW Riley Hospital for Children - Pulmonology, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Health Care d/b/a Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Children's Hospital - Pulmonology, St Louis, Missouri
  - Cohen Children's Medical Center - Lakeville Road, Lake Success, New York
  - Cincinnati Children's Hospital Medical Center - Pulmonology, Cincinnati, Ohio
  - UH Cleveland Medical Center - Pulmonology, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh - Pulmonology, Pittsburgh, Pennsylvania
  - Texas Children's Hospital - Wallace Tower - Pulmonology, Houston, Texas
  - Vermont Lung Center, Colchester, Vermont
  - American Family Childrens Hospital, Madison, Wisconsin
- Australia (4):
  - The Kids Research Institute Australia, Nedlands
  - Women's & Children's Hospital, North Adelaide
  - The Royal Children's Hospital Melbourne, Parkville
  - Children's Health Queensland Hospital and Health Service, South Brisbane
- Canada (2):
  - Hospital for Sick Children - Pulmonology, Toronto
  - British Columbia Children's Hospital, Vancouver
- France (2):
  - Hopital Femme Mere-Enfant, Bron
  - Hopital Necker Enfants Malades - Pulmonology, Paris
- Germany (3):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitatsklinikum Essen, Essen
  - Medizinische Hochschule Hannover - Clinic for Pediatric Pneumology, Allergology and Neonatology, CF-Centre, Hanover
- Sophia Children's Hospital, Rotterdam, Netherlands
- Starship Child Health, Grafton, New Zealand
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset - Göteborg CF-center, Gothenburg
  - Karolinska University Hospital - Pulmonology, Stockholm
- Switzerland (2):
  - Inselspital Bern, Bern
  - Kinderspital Zurich - Abteilung Pneumologie, Zurich
- United Kingdom (2):
  - Noah's Ark Children's Hospital for Wales, Cardiff
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/